CLINICAL TRIAL: NCT00421317
Title: A Phase II Multicentric Trial to Assess Efficacy and Toxicity of Imatinib in Adult Patients With Metastatic Ocular Melanoma
Brief Title: Imatinib in Adult Patients With Metastatic Ocular Melanoma
Acronym: O-Mel-Inib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped at the end of the first step
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Novartis (Industry); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O-Mel-Inib 0508
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Melanoma
Keywords: Ocular, Metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Imatinib — 800 mg/day until disease progression or toxicity

SUMMARY:
The scope of the trial is to determinate the anti-tumoral activity of imatinib in metastatic ocular melanoma patients.

DETAILED DESCRIPTION:
Further study details as provided by Centre Oscar Lambret

ELIGIBILITY:
Inclusion Criteria:

* Metastatic ocular melanoma
* Age > or = 18 years old
* Measurable metastases > or = 10 mm according to RECIST criteria
* PS-WHO < or = 1 or IK > 70 percent
* Normal hepatic function
* PNN > 1500/mm3, platelets > or = 100 000/mm3
* Contraception
* Informed consent signed

Exclusion Criteria:

* Patient with two prior lines of systemic treatment (chemotherapy, immunotherapy or association)
* Other evolutive neoplasic disease
* Severe hepatic insufficiency
* Severe renal insufficiency
* Somatic or psychiatric co-morbidity incompatible with the protocol
* Leptomeningeal or cerebral metastatic dissemination
* Pregnant or lactating woman
* Other antitumoral treatment
* Patient participating to another clinical trial with an experimental drug
* Known hypersensitivity to Imatinib or one of its excipients
* Resecable single metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Progression-free rate at 3 months

SECONDARY OUTCOMES:
Progression-free rate at 6 and 12 months
Response rate according to RECIST criteria
Toxicity
Global survival,Progression-free survival
Predictive genomic factors of response

CONTACTS AND LOCATIONS:
Overall Officials: PENEL Nicolas, MD, Principal Investigator — Centre Oscar Lambret
Locations (12):
- France (12):
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Regional Universitaire, Lille
  - Centre Leon Berard, Lyon
  - Centre Val d'Aurelle Paul Lamarque, Montpellier
  - Institut Curie, Paris
  - Centre Paul Strauss, Strasbourg
  - Hopital Universitaire de Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Gustave Roussy, Villejuif